CLINICAL TRIAL: NCT04489030
Title: Magnifying Narrow-band Imaging for Diagnosis of H. Pylori and Precancerous Gastric Conditions: Comparison With Standard Endoscopy
Brief Title: Magnifying NBI Endoscopy for Gastric Condition
Status: Completed | Type: Observational
Sponsor: Soonchunhyang University Hospital (Other)
Responsible Party: Principal Investigator, Jun-Hyung Cho, Associate Professor, Soonchunhyang University Hospital
Other Study IDs: SCH-NBI endoscopy
Record Dates: First submitted 2020-07-24; First posted 2020-07-28 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Gastritis H Pylori

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen would be obtained for urease test (commercial name: CLOtest) and pathological analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Magnifying narrow-band imaging endoscopy — During endoscopy, gastric mucosal patterns would be examined by magnifying narrow-band imaging.

SUMMARY:
Recently, the improved resolution with standard endoscopy allows the close observation of highly inflamed gastric mucosa without a magnifying view. In a previous study, the investigators established the endoscopic classification of H. pylori-infected stomach by non-magnifying standard endoscopy. One normal RAC pattern and three types of abnormal patterns were observed. Overall diagnostic accuracy for predicting H. pylori-infection was 91.6%. However, there is no comparison study predicting H. pylori-infection and precancerous gastric lesions between standard and magnifying endoscopy.

DETAILED DESCRIPTION:
The investigators aimed to evaluate the diagnostic efficacies of non-magnifying standard endoscopy for predicting H. pylori-infection status and precancerous gastric conditions, compared to magnifying NBI endoscopy

ELIGIBILITY:
Inclusion Criteria:

* Gastroscopy can be performed
* H. pylori test and pathological analysis can be performed

Exclusion Criteria:

* Age < 20 or > 70 years
* Anemia (serum hemoglobin level < 10 g/dL)
* Severe systemic disease
* Advanced chronic liver disease
* Use of certain medications, including proton pump inhibitors, H2- receptor antagonists, or antibiotics
* History of H. pylori eradication
* History of gastric surgery
* Recent history of upper gastrointestinal bleeding

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All of the patients underwent gastroscopy for peptic ulcer, gastric cancer screening in a single academic hospital.
Sampling Method: Non-Probability Sample
Enrollment: 254 (Actual)
Dates: Start 2016-06-01 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
H. pylori infection status | 1 month
  H. pylori positivity would be assessed using rapid urease test.
Degree of chronic gastritis | 1 month
  Gastric atrophy and intestinal metaplasia would be evaluated on the basis of histopathological examination (updated Sydney system).

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Hyung Cho, M.D., Principal Investigator — Digestive Disease Center, Soonchunhyang University Hospital
Locations (1):
- Soonchunhyang University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No